CLINICAL TRIAL: NCT04183478
Title: A Randomized, Double Blinded, Parallel-controlled, Multi-center Phase II/III Study to Compare the Best Support Care (BSC) Plus K-001 Versus BSC Plus Placebo for the Third-line and Later Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: The Efficacy and Safety of K-001 in the Treatment of Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, liwei wang, ONCOLOGY DEPT., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPOG001-05
Record Dates: First submitted 2019-11-25; First posted 2019-12-03 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Tow arms were design in the study. Group 1: Best Support Care (BSC) Plus K-001. Group 2: BSC Plus Placebo. The participants were assign into two groups in a 2:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Support Care Plus K-001 (Experimental): Best support care including analgesic treatment, anti-infection therapy, biliary obstruction treatment, nutritional support, psychological support, reasonable advice from physicians, good communication with patients and etc. K-001 9,720mg per day which means that take K-001 capsule 18 tablets (270mg per tablet) orally twice a day (morning and evening), 56 days as a cycle.
  Interventions: Drug: K-001
- Best Support Care Plus placebo (Placebo Comparator): Best support care is the same as experimental arm. Placebo is take 18 placebo tablets which is the same as K-001 in appearance orally twice a day (morning and evening), 56 days as a cycle.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: K-001 — K-001 is an antitumor active substance (peptidoglycan) which is prepared from the fermentation product of marine microorganism. K-001 is the Chinese first class new drug and get patent licensing in China, America and Japan.
  Arms: Best Support Care Plus K-001
Other: placebo — Placebo which looks the same as K-001 in apparence
  Other Names: K-001 placebo
  Arms: Best Support Care Plus placebo

SUMMARY:
No Standard therapy has been approved for third-line therapy of advanced pancreatic cancer. K001 is peptidoglycan prepared from the marine microorganism, with an anti-tumor activity. Previously, the phase I study of K001 has shown that K001 was safety and had some effectiveness for pancreatic patients. Now, we would like to lunch a randomized, blinded, parallel-controlled, multi-center phase II/III study to compare the best support care (BSC) plus K-001 versus BSC plus placebo for the third-line and later treatment of patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years.
2. Metastatic or locally advanced pancreatic ductal adenocarcinoma which is confirmed by primary and/or metastatic pathology/cytology examination.
3. Had received at least 2 lines chemotherapy regimen, and the disease is progression or the toxicity could not be tolerated.
4. At least 28 days after the last chemotherapy.
5. Had a disease status that was measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST, version1.1).
6. Had an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2.
7. Adequate hepatic, renal, and hematologic functions (neutrophils ≥1.5×10^9/L, platelets ≥ 80×10^9/L,hemoglobin ≥90g/L, total bilirubin within 2.0×the upper limit of normal(ULN), albumin≥30g/L, and ALT and AST≤3×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.5 x ULN and creatinine clearance rate > 30ml/min (Cockcroft-Gault).
8. For women of child-bearing age, the pregnancy test results (serum or urine) within 14 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 60 days post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 60 days post the last administration of study drug.
9. Signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure

Exclusion Criteria:

1. Patients is not confirmed by pathology/cytology examination as pancreatic ductal adenocarcinoma.
2. Target lesions were once treated locally and does not exhibit progression recently.
3. Patients with already diagnosed central nervous system metastasis. Patients with clinical symptoms of central nervous system metastasis should be examined by MRI.
4. Patients with Vater 's ampullary carcinoma or biliary adenocarcinoma.
5. Subject with partial or complete intestinal obstruction,or complete biliary obstruction who are unable to be relieved by active treatment
6. Subject has more than an average of intra-abdominal effusion, or the intra-abdominal effusion could not be control in 2 weeks.
7. Subject has a second malignancy other than curatively resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or other cancers treated with curative intent and no known active disease within 5 years before planned start of study therapy.
8. Female subjects who are pregnant, planning a pregnancy or breast feeding during the study.
9. Subject has an active infection, or a hypertension could not be controlled by drugs, or angina diagnosed within 3 months, or unstable angina pectoris, or myocardial infarction diagnosed within 1 year, or with congestive heart failure (New York Heart Association [NYHA] Class II or III or IV), or with schizophrenia, or with the history of psychotropic substance abuse.
10. Subject has an active infection of hepatitis B (HBV), hepatitis C (HCV) or human immunodeficiency virus (HIV).
11. Subject has received any of the following treatment within the framework of a specific time frame prior to entry:

    1. received operation greater than grade II within 4 weeks;
    2. received extended range radiotherapy within 4 weeks, or locally radiotherapy within 2 weeks;
    3. participated in other therapeutic/interventional clinical trials within 4 weeks;
    4. received locally anti-tumor therapy within 4 weeks；
12. All toxic effects of any prior antitumor therapy resolved to Grade < 2 before the start of study therapy (with the exception of alopecia and pigmentation of skin).
13. Subject has known to be allergic or intolerant to K-001 and its excipients.
14. Other situations that the researchers considered inappropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
overall survival | 6 months after the last subject is enrolled
  The overall survival (OS) of the two groups of FAS was compared. FAS including all the subjects who take at least one dose of the research drug. All the subjects received tumor assessment every 8weeks according to RECIST1.1.

SECONDARY OUTCOMES:
PFS | 6 months after the last subject is enrolled
  All the subjects received tumor assessment every 8weeks according to RECIST1.1 to evaluate the progression-free survival (PFS) .
TTP | 6 months after the last subject is enrolled
  All the subjects received tumor assessment every 8weeks according to RECIST1.1 to evaluate the time to progression (TTP).
ORR | 6 months after the last subject is enrolled
  All the subjects received tumor assessment every 8weeks according to RECIST1.1 to evaluate the objective response rate (ORR).
DCR | 6 months after the last subject is enrolled
  All the subjects received tumor assessment every 8weeks according to RECIST1.1 to evaluate the disease control rate (DCR).
CBR | 6 months after the last subject is enrolled
  According to a questionaire to evaluate the clinical benefit response (CBR) of the two groups.
QOL | 6 months after the last subject is enrolled
  According to a questionaire to evaluate the quality of life (QOL) of the two groups.

OTHER OUTCOMES:
Tumor marker | 6 months after the last subject is enrolled
  blood test to evaluate change of tumor markers, including CEA, CA19-9, CA125, CA724, AFP and etc. of the two groups
Hematology Index | 6 months after the last subject is enrolled
  blood test to evaluate change of D-Dimer, C-Reactive protein (CRP), Albumin (ALB), CAR (CRP/ALB) of the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, Professor, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University; Shukui Qin, Professor, Principal Investigator — Nanjing Bayi Hospital
Locations (1):
- RenJiH, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided